CLINICAL TRIAL: NCT05413031
Title: Treatment of Finger Extensor Tendon Rupture - Comparison Between Static and Relative Motion Splints
Brief Title: Comparing Relative Motion Splint With Static Splint After Hand Extensor Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMB-0110-17
Record Dates: First submitted 2022-06-02; First posted 2022-06-09 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Hand Tendon Injury
MeSH Terms: interventions — Splints

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- relative motion splint (Active Comparator)
  Interventions: Device: relative motion splint
- static splint (Active Comparator)
  Interventions: Device: static splint

INTERVENTIONS:
Device: relative motion splint — splint with ability to move the fingers
  Arms: relative motion splint
Device: static splint — splint with immobility of wrist, and fingers
  Arms: static splint

SUMMARY:
Different splints are used after hand extensor tendon repair (including relative motion splint, static splint, etc.) There is no consensus regarding the benefits of either one.

The aim of this study is to compare clinical outcomes after using different orthoses and rehabilitation methods after hand extensor tendon repair.

Patients are randomly assigned after signing consent to either immobilization with a static splint or a relative motion splint. Patients are examined after 2 and 5 months postoperatively for finger range of motion, grip strength, and DASH questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hand extensor tendon tear in zones 4-7 after surgical repair, that are able to sign a consent form.

Exclusion Criteria:

* patients that did not arrive for a follow-up meeting after 2 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Fingers range of motion | 2 months after surgical repair
  Range of motion in the Metacarpophalangeal joints, Proximal and Distal interphalangeal joints.
Fingers range of motion | 5 months after surgical repair
  Range of motion in the Metacarpophalangeal joints, Proximal and Distal interphalangeal joints.
Grip strength | 2 months after surgical repair
  Measured with the Jamar Hand Dynamometer
Grip strength | 5 months after surgical repair
  Measured with the Jamar Hand Dynamometer
The Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | 2 months after surgical repair
  The scale ranges from 0-to 100 and a higher score interprets as a worse outcome.
The Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | 5 months after surgical repair
  The scale ranges from 0-to 100 and a higher score interprets as a worse outcome.

SECONDARY OUTCOMES:
Fingers range of motion | The change between 2 and 5 months after surgical repair
  Range of motion in the Metacarpophalangeal joints, Proximal and Distal interphalangeal joints.
Grip strength | The change between 2 and 5 months after surgical repair
  Measured with the Jamar Hand Dynamometer
The Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | The change between 2 and 5 months after surgical repair
  The scale ranges from 0-to 100 and a higher score interprets as a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hardy M, Feehan L, Savvides G, Wong J. How controlled motion alters the biophysical properties of musculoskeletal tissue architecture. J Hand Ther. 2023 Apr-Jun;36(2):269-279. doi: 10.1016/j.jht.2022.12.003. Epub 2023 Apr 5. PMID 37029054